CLINICAL TRIAL: NCT02129361
Title: Brief Intervention for Substance Misuse Following Moderate or Severe Traumatic Brain Injury (TBI): A Randomized Controlled Trial
Brief Title: Screening and Brief Intervention for Substance Misuse Following Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Bogner, PhD, ABPP (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jennifer Bogner, PhD, ABPP, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012H0424
Record Dates: First submitted 2014-04-28; First posted 2014-05-02 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Crisis Intervention; Mass Screening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adapted Screening and Brief Intervention (Experimental): Adapted Screening and Brief Intervention: Participants will be screened for substance use, receive education regarding the effects of substance misuse, participate in a motivation interview, and participate in a booster session one month later
  Interventions: Behavioral: Adapted Screening and Brief Intervention (Adapted SBI)
- Screening & Education Attention Control (Active Comparator): Screening & Education Attention Control: Participants will be screened for substance use, receive education regarding the effects of substance misuse, and participate in a booster session one month later
  Interventions: Behavioral: Screening & Education Attention Control

INTERVENTIONS:
Behavioral: Adapted Screening and Brief Intervention (Adapted SBI)
  Arms: Adapted Screening and Brief Intervention
Behavioral: Screening & Education Attention Control
  Arms: Screening & Education Attention Control

SUMMARY:
This study is investigating one way to improve health and healthy habits after traumatic brain injury (TBI). The primary goal of this study is to determine if a brief intervention accommodated for persons with moderate or severe TBI is effective in reducing alcohol misuse during the year following injury. It is hypothesized that an adapted Screening, Education and Brief Intervention (adapted SBI) will reduce the number of alcoholic drinks consumed per week over the year following discharge from inpatient rehabilitation, in comparison to a Screening and Education Attention Control condition (SEA control).

ELIGIBILITY:
Inclusion Criteria:

* Sustained a TBI, defined as damage to brain tissue caused by external force and evidenced by loss of consciousness, post-traumatic amnesia, skull fracture, or objective neurological findings
* History of alcohol misuse within the year prior to injury
* Be at least 18 years old
* English-speaking
* Have cleared post-traumatic amnesia
* Able and willing to provide informed consent

Exclusion Criteria:

* Language impairments that would preclude participation in interview
* Has not cleared post-traumatic amnesia before discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2014-03; Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Number of alcoholic drinks consumed per week in past month | Change from baseline to 12 months post-discharge
  Number of drinks will be recorded at baseline, 6, 9, and 12 months. We will be measuring change in the number of drinks consumed of the course of the year, with the primary outcome being measured at the 12 month assessment.

SECONDARY OUTCOMES:
Frequency of alcohol binges in past month | Change in the number of alcohol binges baseline to 12 months post-discharge
  Binge is defined as 4 or more drinks in a day for women, 5 or more drinks in a day for men
Alcohol expectancies | 12 months post-discharge
  Measured by the shortened Alcohol Expectancies Questionnaire-III
Number of facts retained about negative consequences of substance misuse | 12 months post-discharge
  Count of number of facts, maximum=8
Number of alcoholic drinks consumed per week during the past month | Change from baseline to 3 months post-discharge
  Count of number of facts, maximum=8
Number of alcoholic drinks consumed per week in the past month | Change from baseline to 6 months post-discharge
Frequency of alcohol binges in past month | Change from baseline to 6 months post-discharge
  Binge is defined as 4 or more drinks in a day for women, 5 or more drinks in a day for men
Number of alcohol binges in past month | Change from baseline to 3 months post-discharge
  Binge is defined as 4 or more drinks in a day for women, 5 or more drinks in a day for men
Alcohol expectancies | 6 months post-discharge
  Measured by the shortened Alcohol Expectancies Questionnaire-III
Alcohol expectancies | 3 months post-discharge
  Measured by the shortened Alcohol Expectancies Questionnaire-III
Number of facts retained about negative consequences of alcohol use | 3 months post-discharge
  Count of number of facts, maximum=8
Number of facts retained about negative consequences of alcohol use | 6 months post-discharge
  Count of number of facts, maximum=8

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Bogner, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Bogner J, Corrigan JD, Peng J, Kane C, Coxe K. Comparative effectiveness of a brief intervention for alcohol misuse following traumatic brain injury: A randomized controlled trial. Rehabil Psychol. 2021 Nov;66(4):345-355. doi: 10.1037/rep0000405. Epub 2021 Oct 7. PMID 34618511